CLINICAL TRIAL: NCT01705457
Title: Impact of Vitamin A Supplementation on RAR Gene Expression in PBMC Cells in Multiple Sclerotic Patients
Brief Title: Impact of Vitamin A on RAR Gene Expression in Multiple Sclerosis
Acronym: RAR
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 91-03-161-19476
Record Dates: First submitted 2012-10-09; First posted 2012-10-12 (Estimated); Last update posted 2012-10-12 (Estimated); Status verified 2012-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: multiple sclerosis; Vitamin A; retinoic acid receptor; retinoic x receptor
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — retinol palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- with Multiple Sclerosis, vitamin A (Active Comparator): Patients with Multiple Sclerosis confirmed Relapsing Remitting Type
  Interventions: Drug: Dietary Supplement: vitamin A
- with multiple sclerosis,placebo (Placebo Comparator): Patients with Multiple Sclerosis confirmed Relapsing Remitting Type
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dietary Supplement: vitamin A — 25000 IU/day vitamin A for 6 months
  1 Cap/Day
  1 cap placebo/day for 6 month
  Other Names: Retinyl palmitate
  Arms: with Multiple Sclerosis, vitamin A
Drug: placebo
  Arms: with multiple sclerosis,placebo

SUMMARY:
The aim of this study is the comparison between the effects of supplementation with 25000 IU preformed vitamin A (retinyl palmitate)on retinoic acid receptor and retinoic x receptor expression.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic inflammatory disease where Th1 like responses from myelin-specific CD4+ T cells, as secretion of pro-inflammatory IFNγ, are believed to play a major role in the pathogenesis. The myelin-specific T cells that mediate tissue destruction in MS are believed to become activated outside the central nervous system (CNS) in lymphoid tissue and when they cross the blood brain barrier they will re-encounter their antigen. Immune deviation is the redirection of the immune response from most often Th1 like responses to Th2 like responses, even though the opposite can also occur. Vitamin A or Vitamin A-like analogs known as retinoids, are potent hormonal modifiers of type 1 or type 2 responses but a definitive description of their mechanism(s) of action is lacking. High level dietary vitamin A enhances Th2 cytokine production and IgA responses, and is likely to decrease Th1 cytokine production. Retinoic acid(RA) inhibits IL12 production in activated macrophages, and RA pretreatment of macrophages reduces IFNγ production and increases IL4 production in antigen primed CD4 T cells. Supplemental treatment with vitamin A or RA decreases IFNγ and increases IL5, IL10, and IL4 production by increase of retinoic acid receptor and retinoic x receptor .

Record Verification Date: August 2011

ELIGIBILITY:
Inclusion Criteria:

* Patients who have used interferon beta in last 3 months.
* Patients with 0-5 EDSS

Exclusion Criteria:

* Patients who have diseases which affect on Th1/Th2 balance such as asthma, active viral infections, and autoimmune diseases, OR
* Patients who have allergy to vitamin A compounds, OR
* Patients who have used vitamin supplements in last 3 months.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-02; Primary Completion 2013-02 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Gene expression of RAR(Relative quantification) | Change from baseline at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ali Akbar saboor Yaraghi, PhD, Study Chair — Tehran University of Medical Sciences; Sama Bitarafan, MD, PhD student, Principal Investigator — Tehran University of Medical Siences
Locations (1):
- Tehran University of Medical Sciences,, Tehran, Iran